CLINICAL TRIAL: NCT00275535
Title: A Prospective, Randomized Trial of Calcineurin-Inhibitor Withdrawal in Renal Allograft Recipients
Brief Title: The Comparison of Tacrolimus and Sirolimus Immunosuppression Based Drug Regimens in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Genzyme, a Sanofi Company (Industry); Roche Pharma AG (Industry)
Responsible Party: Mark D. Stegall, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 124-01
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Kidney Diseases
Keywords: kidney transplantation; immunosuppression; calcineurin inhibitor; sirolimus; chronic allograft nephropathy
MeSH Terms: conditions — Kidney Diseases | interventions — Antilymphocyte Serum; thymoglobulin; Mycophenolic Acid; Prednisone; Tacrolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): Calcineurin inhibitor arm, consisting of treatment with tacrolimus, mycophenolate mofetil, and prednisone.
  Interventions: Drug: Anti-thymocyte globulin; Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Tacrolimus
- Sirolimus (Active Comparator): Calcineurin inhibitor-free arm, consisting of treatment with rapamycin, mycophenolate mofetil, and prednisone.
  Interventions: Drug: Anti-thymocyte globulin; Drug: Mycophenolate mofetil; Drug: Prednisone; Drug: Sirolimus

INTERVENTIONS:
Drug: Anti-thymocyte globulin — Thymoglobulin 1.5 mg/kg/d (days 0,1,2,4,6)
  Other Names: Thymoglobulin; Atgam
Drug: Mycophenolate mofetil — Mycophenolate mofetil 750 mg p.o. b.i.d.- maintenance
  Other Names: CellCept
Drug: Prednisone — Prednisone 500 mg/day initially, tapered to 5 mg/day by day 92
  Other Names: Deltasone; Liquid Pred; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred; Sterapred DS
Drug: Tacrolimus — Tacrolimus - maintain trough levels of 6-8 ng/ml (whole blood Imx assay)
  Other Names: Prograf; Advagraf; Protopic
  Arms: Tacrolimus
Drug: Sirolimus — Rapamycin 3 to 5 mg/day; adjust to the high-performance liquid chromatography (HPLC) blood level 15 to 20 ng ml
  Other Names: Rapamune
  Arms: Sirolimus

SUMMARY:
This study was done to find out which treatment, tacrolimus or sirolimus, leads to better long-term kidney function in kidney transplant patients.

DETAILED DESCRIPTION:
The aim of this study was to compare the complete avoidance of calcineurin inhibitors (CI) using a sirolimus-based immunosuppressive regimen to a tacrolimus-based regimen in kidney transplantation. This study was a prospective open-label trial randomizing patients to receive tacrolimus, mycophenolate mofetil and prednisone or sirolimus, mycophenolate mofetil and prednisone. All patients received antithymocyte globulin induction. All rejection episodes were proven by biopsy. The hypothesis was that CI free immunosuppression after kidney transplantation will lead to an increase in glomerular filtration rate (GFR) at one year after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Living and deceased donor kidney transplant recipients at the Mayo Clinic, Rochester, Minnesota

Exclusion Criteria:

* Patients with type 1 diabetes less than 50 years of age who receive a living donor kidney transplant followed by a pancreas transplant
* Pediatric patients (<18 years of age)
* Multi-organ transplants (e.g., kidney-pancreas, kidney-liver)
* ABO-incompatible or positive crossmatch recipients (ABO incompatibility is an immune system reaction that occurs when blood from two different and incompatible blood types are mixed together.)
* Patients with severe hyperlipidemia (serum cholesterol >350 mg/dl or serum triglycerides >500 mg/dl
* Patients with severe leukopenia (White Blood Cell count [WBC]<3000 10^3/ml)
* Patients unwilling to return to the transplant center for late follow-up visits
* Body mass index (BMI) ≥ 32 with incisional problems post transplant (as determined by renal transplant surgeon

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2001-04; Primary Completion 2007-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) (iothalamate clearance) at 12 months following transplantation | 12 months following transplantation
  Glomerular filtration rate (Iothalamate clearance) at 12 months following transplantation.

SECONDARY OUTCOMES:
GFR (iothalamate clearance) at other time points | 24 months
Other measures of renal function (serum creatinine, proteinuria and albuminuria) | 24 months
Acute rejection both early and after tacrolimus withdrawal | 24 months
Patient and graft survival | 24 months after transplantation
Complications-especially hypertension, diabetes, dyslipidemia | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Dean PG, Grande JP, Sethi S, Park WD, Griffin MD, Cosio FG, Larson TS, Stegall MD. Kidney transplant histology after one year of continuous therapy with sirolimus compared with tacrolimus. Transplantation. 2008 Apr 27;85(8):1212-5. doi: 10.1097/TP.0b013e31816a8ae6. PMID 18431244
- [Result] Larson TS, Dean PG, Stegall MD, Griffin MD, Textor SC, Schwab TR, Gloor JM, Cosio FG, Lund WJ, Kremers WK, Nyberg SL, Ishitani MB, Prieto M, Velosa JA. Complete avoidance of calcineurin inhibitors in renal transplantation: a randomized trial comparing sirolimus and tacrolimus. Am J Transplant. 2006 Mar;6(3):514-22. doi: 10.1111/j.1600-6143.2005.01177.x. PMID 16468960